CLINICAL TRIAL: NCT05850494
Title: Randomized, DB, Crossover Study to Assess Bronchospasm Potentially Induced by HFO MDI vs. HFA MDI Propellant in Participants With Asthma Well/Partially Controlled on SABA With or Without Low-Dose ICS
Brief Title: Study to Assess Bronchospasm Potentially Induced by Next-Generation Propellant vs HFA Propellant in an MDI in Participants With Well/Partially Controlled Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5985C00007
Record Dates: First submitted 2023-04-28; First posted 2023-05-09 (Actual); Results first posted 2025-07-30 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-11

CONDITIONS: Asthma
Keywords: Asthma, Bronchospasm
MeSH Terms: conditions — Asthma; Bronchial Spasm

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to assess bronchospasm potentially induced by hydrofluoroolefin (HFO) metered dose inhaler (MDI) as compared with hydrofluoroalkane (HFA) MDI in participants with asthma, well controlled or partially controlled on treatment for asthma, including, low-dose inhaled corticosteroid (ICS) daily or low-dose ICS/formoterol as needed (not approved in the US), or short-acting beta2-agonists (SABA) as needed, or low-dose ICS whenever SABA as needed is used.
  Study details include:
  * The study duration will be up to 37 days.
  * The treatment duration will be 1 day for each treatment period.
  * The visit frequency will be approximately every 1 week.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is double blinded with regard to treatment (MDI administered with 2 different propellants [Treatment A or B]), ie, the sponsor, the investigator, all clinical staff involved in the clinical study, the participants, and the study monitor will remain blinded, unless safety concerns or a regulatory requirement necessitate unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: HFO propellant only MDI (Experimental): Test arm, 4 inhalations per dose
  Interventions: Drug: HFO MDI
- Treatment B: HFA propellant only MDI (Active Comparator): Reference arm, 4 inhalations per dose
  Interventions: Drug: HFA MDI

INTERVENTIONS:
Drug: HFA MDI — * Dose formulation: MDI
  * Unit dose strength(s): Reference (propellant only)
  * Dosage Level: 4 inhalations, single dose
  * Route of administration: Oral inhalation
  * Participants will receive treatment A in 1 or 2 possible sequences AB or BA
  Other Names: Propellant in MDI
  Arms: Treatment B: HFA propellant only MDI
Drug: HFO MDI — * Dose formulation: MDI
  * Unit dose strength(s): Experimental (propellant only)
  * Dosage Level: 4 inhalations, single dose
  * Route of administration: Oral inhalation
  * Participants will receive treatment A in 1 or 2 possible sequences AB or BA
  Other Names: Propellant in MDI
  Arms: Treatment A: HFO propellant only MDI

SUMMARY:
A study to assess bronchospasm potentially induced by HFO MDI as compared with HFA MDI in participants with well controlled or partially controlled asthma

DETAILED DESCRIPTION:
This is a phase 3b, multicentre, randomized, double-blind, single-dose crossover study comparing the safety and tolerability of HFO MDI with HFA MDI delivered in participants with well controlled or partially controlled asthma defined as an ACQ-5 score < 1.5.Eligible participants are at least 18 years of age and no older than 45 years of age and are required to have asthma as defined by GINA guidelines (GINA 2022). Participants are required to be well controlled or partially controlled on their current treatment for asthma, including, low-dose ICS daily or low-dose ICS/formoterol as needed (not approved in the US), or SABA as needed, or low-dose ICS whenever SABA as needed is used. The primary objective is to assess the potential change in FEV1 induced by HFO MDI as compared with HFA MDI in participants with asthma.

This study will be conducted at approximately 5 sites in the US and will randomize approximately 52 adult participants to achieve 46 completers.

The study will be conducted for a maximal 37 days and will comprise:

* A screening period approximately 14 (±2) days prior to first dosing
* Two treatment periods of 1 day each, with a 3 to 12-day washout period between the 2 treatment periods
* A final safety follow-up visit via telephone contact 3 to 7 days after the final dose administration in Treatment Period 2

Single dose study treatment will be administered via MDI device as 4 inhalations:

* Treatment A: HFO propellant only MDI; 4 inhalations per dose - test formulation
* Treatment B: HFA propellant only MDI; 4 inhalations per dose - reference formulation

ELIGIBILITY:
Inclusion Criteria:

* Age

  1. Male and female participant must be 18 to 45 years of age inclusive, at the time of signing the informed consent form (ICF).

     Type of Participant and Disease Characteristics
  2. Participants who have a documented history of physician-diagnosed asthma

     ≥ 12 months prior to Visit 1, according to GINA guidelines (GINA 2022).
  3. Participants who are well controlled or partially controlled on their current treatment for asthma, including, low-dose ICS daily or low-dose ICS/formoterol as needed (not approved in the US), or SABA as needed, or low-dose ICS whenever SABA as needed is used (low-dose ICS as defined by GINA 2022 in Table 4), for 4 weeks prior to screening.
  4. ACQ-5 total score < 1.5 at Visit 1.
  5. A pre-bronchodilator FEV1 > 60% predicted normal value at Visit 1.
  6. Demonstrate acceptable MDI administration technique.

     Sex and Contraceptive/Barrier Requirements
  7. Females must be not of childbearing potential, or should be using a form of highly effective birth control as defined below:
* Female participants Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women included in this study will be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatment and follicle-stimulating hormone levels in the postmenopausal range.
* Female participants of childbearing potential must use one highly effective form of birth control. A highly effective method of contraception is defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly. At enrolment, women of childbearing potential who are sexually active with a non-sterilized male partner should be stable on their chosen method of highly effective birth control, as defined below, and willing to remain on the birth control until at least 14 days after last dose of study intervention. Cessation of contraception after this point should be discussed with a responsible physician.

Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together. All women of childbearing potential must have a negative serum pregnancy test result at Visit 1.

* Highly effective birth control methods are listed below:
* Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant (defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of exposure to study intervention, and withdrawal are not acceptable methods of contraception.
* Contraceptive subdermal implant
* Intrauterine device or intrauterine system
* Oral contraceptive (combined or progesterone only)
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Male partner sterilization with documentation of azoospermia prior to the female participant's entry into the study, and this male is the sole partner for that participant. The documentation on male sterility can come from the site personnel's review of participant's medical records, medical examination and/or semen analysis or medical history interview provided by her or her partner.
* Bilateral tubal ligation Informed Consent 8 Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* Medical Conditions

  1. Life-threatening asthma defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s).
  2. Current smokers, former smokers with > 10 pack-years history, or former smokers who stopped smoking < 6 months prior to Visit 1 (including all forms of tobacco, e-cigarettes or other vaping devices, and marijuana).
  3. Historical or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neurological, endocrine, gastrointestinal, or pulmonary (e.g., active tuberculosis, bronchiectasis, pulmonary eosinophilic syndromes, COPD, and uncontrolled severe asthma). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the participant at risk through participation, or that could affect the safety/tolerability analysis.
  4. Any respiratory infection or asthma exacerbation treated with systemic corticosteroids and/or additional ICS treatment in the 8 weeks prior to Visit 1 and throughout the screening period.
  5. Hospitalization for asthma within 1 year prior to Visit 1.
  6. Admission to intensive care unit or mechanical ventilation due to asthma exacerbation.
  7. Known history of drug or alcohol abuse within 12 months of Visit 1.

     Prior/Concomitant Therapy
  8. Do not meet the stable dosing period prior to Visit 1 (see Table 5) or unable to abstain from protocol-defined prohibited medications during screening and treatment periods (see Table 6 and Table 7).
  9. Receipt of COVID-19 vaccine (regardless of vaccine delivery platform, e.g., vector, lipid nanoparticle) ≤ 7 days prior to Visit 1 (from last vaccination or booster dose).

Prior/Concurrent Clinical Study Experience 10 Participation in another clinical study with an investigational product administered within 30 days or 5 half-lives (whichever is longer). 11 Participants with a known hypersensitivity to HFO or HFA or any of the excipients of the product. 12 Previously randomized into a study with an HFO-containing MDI.

Diagnostic Assessments 13 Any clinically relevant abnormal findings in physical examination, clinical chemistry, hematology, urinalysis, vital signs, or electrocardiogram (ECG), which in the opinion of the investigator, may put the participant at risk because of his/her participation in the study. Note: Participants with ECG QT interval corrected for heart rate using Fridericia's formula (QTcF) > 480 msec will be excluded. Participants with high degree atrioventricular block II or III, or with sinus node dysfunction with clinically significant pauses who are not treated with pacemaker will also be excluded.

Other Exclusions 14 Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site). 15 Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

16 Previous enrolment or randomisation in the present study. 17 For women only - currently pregnant (confirmed with positive pregnancy test), breast feeding, or planned pregnancy during the study or women of childbearing potential not using acceptable contraception measures. 18 Study investigators, sub-investigators, coordinators, and their employees or immediate family members.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, Principal Investigator — Northeast Medical Research Associates, Inc.; Craig LaForce, MD, Principal Investigator — North Carolina Clinical Research; Allen T Funkhouser, MC, Principal Investigator — EPIMRD Inc.; Jeffrey Tillinghast, MD, Principal Investigator — The Clinical Research Center, LLC.
Locations (4):
- United States (4):
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, El Paso, Texas

REFERENCES:
- [Result] Buhl R, Tanase AM, Hosoe M, Cao W, Demin I, Bartels C, Jauernig J, Ziegler D, Patalano F, Hederer B, Kanniess F, Tillmann HC. A randomized, double-blind study to compare the efficacy and safety of two doses of mometasone furoate delivered via Breezhaler(R) or Twisthaler(R) in patients with asthma. Pulm Pharmacol Ther. 2020 Jun;62:101919. doi: 10.1016/j.pupt.2020.101919. Epub 2020 May 7. PMID 32387408
- [Result] Global Initiative for Asthma (GINA). Global Strategy for Asthma Management and Prevention, 2022. http://ginasthma.org.
- [Result] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Result] Investigator's Brochure - Budesonide, Glycopyrronium and Formoterol Fumarate Inhalation Aerosol (BGF MDI); Budesonide and Formoterol Fumarate Inhalation Aerosol (BFF MDI); Budesonide Inhalation Aerosol (BD MDI); Glycopyrronium Inhalation Aerosol (GP MDI) (Also known as PT010 [BGF MDI], PT009 [BFF MDI], PT008 (BD MDI); PT001 (GP MDI); Edition Number 9.0, 16 September 2022.
- [Result] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Result] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Result] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Result] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Result] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Derived] Pleasants RA, Bell AS, Jassal M, Xu J, Petullo D, Raphiou I, Aurivillius M, Bondarov P, Patel M. A Randomized, Double-Blind Crossover Study of Change in Post-Dose Lung Function with Hydrofluoroolefin-1234ze, a Next-Generation Propellant for Metered Dose Inhalers, in Participants with Asthma. J Aerosol Med Pulm Drug Deliv. 2025 Oct;38(5):275-283. doi: 10.1089/jamp.2024.0061. Epub 2025 Jun 24. PMID 40551410
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5985C00007&attachmentIdentifier=ee73a15b-ba47-453b-b020-74fcd162e7a8&fileName=d5985c00007-synopsis-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence HFA-HFO: HFA propellant only metered-dose inhaler (4 inhalations per dose - reference formulation) then HFO propellant only metered-dose inhaler (4 inhalations per dose - test formulation)
- Sequence HFO-HFA: HFO propellant only metered-dose inhaler (4 inhalations per dose - test formulation) then HFA propellant only metered-dose inhaler (4 inhalations per dose - reference formulation)
Period: Overall Study
Arm/Group | Sequence HFA-HFO | Sequence HFO-HFA
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence HFO-HFA | Sequence HFA-HFO | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (9.78) | 30.9 (7.86) | 32.4 (8.90)
Age, Customized [Number; unit: Participants] — Age at Screening Population: Full Analysis Set
  Participants
    18-45 | 26 | 26 | 52
    Missing | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Full Analysis Set
  Participants
    Female | 17 | 19 | 36
    Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Full Analysis Set
  Participants
    Hispanic or Latino | 8 | 7 | 15
    Not Hispanic or Latino | 18 | 19 | 37
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Full Analysis Set
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 4 | 7
    White | 22 | 21 | 43
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Country [Count of Participants; unit: Participants] — Full Analysis Set
  Participants
    USA | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve From 0 to 15 Minutes (AUC0-15 Min) Post-dose
Description: The change from baseline (30 minutes pre-dose) in normalized FEV1 AUC0-15 min postdose induced by Treatment HFO was compared with Treatment HFA.
Time Frame: 30 minutes prior to dosing and at 5, 15, and 30 minutes post-dose
Population: Primary Analysis Set
Measure: Mean (Standard Deviation); unit: Litres
Groups:
- Treatment HFO: HFO propellant only metered-dose inhaler; 4 inhalations per dose - test formulation
- Treatment HFA: HFA propellant only metered-dose inhaler; 4 inhalations per dose - reference formulation
Arm/Group | Treatment HFO | Treatment HFA
Number analyzed (Participants) | 52 | 52
Litres
  Baseline FEV1 (30 minutes pre-dose) | 2.969 (0.6660) | 2.970 (0.6463)
  Normalized FEV1 AUC0-15 min | 2.955 (0.6577) | 2.965 (0.6474)
  Change from baseline in normalized FEV1 AUC0-15 min post-dose | -0.014 (0.0794) | -0.004 (0.0565)
Statistical Analysis 1: Comparison: Treatment HFO vs Treatment HFA; Test type: Non-Inferiority — Non-inferiority margin of -0.200 L at a one-sided significance level of 0.025; Mixed Models Analysis — P-Value not applicable since a non-inferiority test was used for the analysis; Mean Difference (Net) = -0.009, 95% CI 2-sided [-0.037 to 0.018], Standard Error of Mean 0.0136

2. Secondary Outcome: Number of Participants With Bronchospasm Events
Description: The potential of Treatment HFO to induce bronchospasm was compared with Treatment HFA. The number of participants with bronchospasm events post-dose (5 or 15 minutes post-dose) from baseline (30 minutes pre-dose) for each treatment is presented.
  An event of bronchospasm is defined as a reduction in FEV1 of >15% from baseline (i.e. the FEV1 value obtained within 30 minutes prior to study intervention administration) at 5 or 15 minutes post-dose, with associated symptoms of wheezing, shortness of breath, or cough.
Time Frame: 30 minutes prior to dosing and at 5 and 15 minutes post-dose
Population: Safety Set
Measure: Number; unit: Participants
Arm/Group | Treatment HFO | Treatment HFA
Number analyzed (Participants) | 52 | 52
Participants | 0 [NC to NC] | 0 [NC to NC]

3. Secondary Outcome: Safety and Tolerability Evaluated in Terms of Adverse Events (AEs)
Description: The number of AEs, SAEs, and AESIs for Treatment HFO and Treatment HFA are presented.
Time Frame: From screening (Day - 14) to the last dose (day 8) + 7 days
Population: Safety Set
Measure: Number; unit: Events
Arm/Group | Treatment HFO | Treatment HFA
Number analyzed (Participants) | 52 | 52
Events
  Any AE | 2 | 4
  Serious AE (SAE) | 0 | 0
  Any SAE with outcome death | 0 | 0
  Any AE leading to discontinuation of investigational product | 0 | 0
  Any possibly related AE | 1 | 0
  Any possibly related SAE | 0 | 0
  Any AE of special interest | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events with start date on or after the date of treatment during treatment period 1 up to (and including) 7 days after the last dose date were included, up to 20 days.
Description: Subjects with multiple occurrences in the same category are counted once per category regardless of the number of occurrences.
Arm/Group | Treatment HFO | Treatment HFA
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 2/52 | 2/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment HFO (N=52) | Treatment HFA (N=52)
Fatigue (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator shall be entitled to publish the results of, or make presentations related to, the Study, provided that any publications or presentations to be made within 2 years after completion of the Study shall require the Sponsor's prior written consent.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT05850494/Prot_002.pdf
  • Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT05850494/SAP_001.pdf